CLINICAL TRIAL: NCT04662164
Title: A Randomized, Double-blind, Placebo-Controlled, Repeat-Dose Study to Assess the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of L47 in Subjects With Type 2 Diabetes Mellitus on Stable Metformin
Brief Title: A Study to Access the Efficacy in Type 2 Diabetes Mellitus on Stable Metformin
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not approved by CFDA
Sponsor: Shanghai HEP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: L47-DM-II-01
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes Patients
Keywords: hepalatide; FBG; TG; TC; PK

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo (Placebo Comparator): control
  Interventions: Drug: hepalatide
- 4.2mg hepalatide (Active Comparator): low dose
  Interventions: Drug: hepalatide
- 6.3mg hepalatide (Active Comparator): middle dose
  Interventions: Drug: hepalatide
- 8.4mg hepalatide (Active Comparator): high dose
  Interventions: Drug: hepalatide

INTERVENTIONS:
Drug: hepalatide — 3 different dosage will be given sequentially to T2D patients
  Other Names: L47

SUMMARY:
This is a randomized, double-blind, placebo-controlled, repeat-dose study to evaluate the safety, tolerability, PK, and PD of L47 as an add-on treatment to stable metformin therapy in patients with T2DM. Approximately 30 subjects will be randomized into the study at up to two investigational sites. The study includes a screening period of up to 28 days, with a three-day, single-blind, placebo lead-in period; a four-week, double-blind treatment period; and a one-week follow-up period. There will be 2 inpatient stays (Day -3 to 2 and 27 to 29) and daily outpatient visits during treatment period. During the follow-up period, there will be 1 outpatient visit at the end of the study. There will be 3 cohorts of 10 subjects each to be enrolled sequentially. In each cohort, subjects will be randomized in a 4:1 ratio to receive either L47 or placebo subcutaneously. Subjects will monitor fasting capillary glucose (finger sticks or self-monitoring of blood glucose, SMBG) during the lead-in, treatment, and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have received a diagnosis of T2DM ≥3 months prior to screening
2. Subjects who have taken a stable metformin dose for at least one month prior to screening and are not currently taking other anti-diabetic drugs
3. Males or females between 18 and 70 years of age, inclusive. Females must have agreed to use appropriate birth control throughout the study or be surgically sterile (hysterectomy, tubal ligation, bilateral oophorectomy) or post-menopausal for 1 year (with follicle stimulating hormone in menopausal range). A serum pregnancy test was performed for women of childbearing potential at the screening visit and at Day -1.
4. Male patients with sexual partners of childbearing potential and female patients of childbearing potential must have agreed to use 1 of the following contraception methods:

   * One form of barrier method contraception (eg, latex condom with spermicide or a diaphragm with intravaginal spermicide or cervical cap with spermicide) in addition to a male patient's female partner(s) taking an oral contraceptive; or
   * Two forms of barrier method contraception (eg, latex condom with spermicide AND a diaphragm with intravaginal spermicide or cervical cap with spermicide);
5. Subjects who have a body mass index ≥19 kg/m2 and ≤35 kg/m2
6. Subjects who have a Hemoglobin A1c(HBA1c) ≥6.5% and ≤10.5%, as assessed by the central laboratory
7. Current non-smokers who have not used tobacco or nicotine in any form at least 6 months prior to dosing
8. Currently have not used nicotine and non-nicotine vaping/electronic cigarette products in the last 6 months
9. Fasting plasma glucose >110 mg/dL and <240 mg/dL;
10. Willing and able to be confined to the investigational site as required by the protocol;
11. Willing and able to comply with the investigational nature of the study and able to communicate well with the Principal Investigator and clinical staff; and
12. Able to comprehend and willing to provide written informed consent in accordance with institutional and regulatory guidelines.

Exclusion Criteria:

1. Have a condition that is a contraindication for use of metformin per Label at screening or at baseline visit;
2. History of type 1 diabetes mellitus, or latent autoimmune diabetes in adults, diabetic neuropathy, retinopathy or nephropathy
3. History of renal transplantation or are receiving renal dialysis at the time of screening
4. History of severe symptomatic hypoglycemia within six months of screening
5. History of diabetic ketoacidosis or other types of metabolic acidosis
6. History of diabetic gastroparesis
7. History of chronic or acute pancreatitis
8. History of hemochromatosis
9. History or presence of clinically significant cardiovascular disease (including a history of unstable angina, acute myocardial infarction, coronary artery bypass graft, percutaneous coronary intervention, or New York Heart Association Class III or IV congestive heart failure within six months prior to screening)
10. Uncontrolled hypertriglycerides >500 mg/dL
11. History of acute or chronic renal disease; estimated glomerular filtration rate (eGFR) ≤60 ml/min/1.73m2
12. Inability to tolerate subcutaneous injections
13. History of allergy, sensitivity or intolerance to peptide products or history of severe hypersensitivity to drugs, foods or other environmental allergens
14. History of coagulation disorders with a potential of causing excessive bleeding or a history of unexplained excessive bleeding
15. Use of warfarin or other anti-coagulation drugs. The use of anti-platelet drugs such as acetylsalicylic acid (daily use) and/or clopidogrel that are prescribed for prevention of cardiovascular events is permitted.
16. Use of systemic glucocorticoids within two weeks of the screening visit, including oral or injectable, or planned use of intermittent systemic corticosteroids during the course of the study. The use of inhaled or topical corticosteroids is permitted.
17. Inadequate venous access
18. Heart rate (HR) <40 bpm or >100 bpm at screening
19. Any clinically significant ECG abnormality at screening (as deemed by the Investigator) including: second or third degree AV block, sick sinus syndrome, atrial fibrillation, presence of other significant dysrhythmias, prolonged QTcF interval >450 msec (the average value for the triplicate ECG at screening and check-In), or history of prolonged QT syndrome

    Note: The following are ECG findings considered not clinically significant without consulting the Medical Monitor:
    * Mild first-degree atrioventricular block (PR interval <0.23 sec)
    * Right or left axis deviation
    * Incomplete right bundle branch block
    * Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic subjects
20. Reported history of liver disease and/or liver enzymes (alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyltransferase (GGT), total bilirubin >2 times the upper limit of normal (ULN) on screening
21. Reported history of clinically significant cerebrovascular or neurological disease including transient ischemic attack, stroke, seizure disorder within one year prior to screening
22. Psychiatric disease including major depression, bipolar disorder, anxiety, or schizophrenia, or other medical condition that, in the opinion of the Investigator, would interfere with the evaluation of study drug safety
23. Use of weight loss medication at screening or prior weight loss surgery involving the gastrointestinal tract
24. Has active or untreated malignancy or has been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer, or in situ carcinomas of the cervix or prostate) for <5 years
25. History of alcoholism or drug abuse within two years prior to dosing

    - Typical weekly alcohol consumption of ≥ 14 alcoholic drinks. One drink is defined as one can of beer (12 oz, approximately 330 mL 5% alcohol), one glass of wine (5 oz, approximately 140 mL 12% alcohol), or one shot of liquor (1.5 oz, approximately 40 mL 40% alcohol)
26. History of acquired immune deficiency syndrome, hepatitis C, or positive test at screening for human immunodeficiency virus antibody, hepatitis B surface antigen, or hepatitis C antibody
27. Patients with a history of blood loss (including blood donation) estimated to be >450 mL within 56 days (or ≥200 mL within 1 month) prior to the Screening Visit
28. Use of any herbal medications or vitamins from the Screening Visit throughout the duration of the study
29. Use of drugs including angiotensin II receptor antagonists (sartans), hydroxymethylglutaryl coenzyme A reductase inhibitors (statins), angiotensin converting enzyme inhibitors (prils) and hypoglycemic drugs (glinides) , other important drugs using OATP1B1/OATP1B3 as main transporters, and other important drugs with NTCP inhibition (appendix 3);
30. Use of another investigational drug or device within 60 days prior to receiving the first dose of study drug in this study, or within five half-lives of the previous investigational drug, whichever is longer
31. Investigational site personnel directly affiliated with this study and/or their immediate families. Immediate family was defined as a spouse, parent, child, or sibling, whether biological or legally adopted
32. Poor mental function or any other reason to expect subject's difficulty in complying with the requirements of the study
33. History or presence of any medical condition or disease, including known alcohol or drug abuse, which, in the opinion of the Investigator, could have interfered with the conduct of the study or would have put the patient at unacceptable risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
24-hour weighed mean glucose (WMG) | 28 days
  The change from baseline in the 24-hour WMG calculated is as the AUC0-24h divided by 24 using linear trapezoidal method. [Time frame: Baseline (Day -1), to Day 28]
AEs | 28 days
  Number and percentage of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), number of subjects discontinuing due to AEs

SECONDARY OUTCOMES:
fasting plasma glucose | 28 days
  Change from baseline in fasting plasma glucose (FPG) level [Time frame: Baseline (Day -1), Day28]

IPD SHARING:
Plan to Share IPD: No